CLINICAL TRIAL: NCT05895617
Title: Is the Occuity Pachymeter Non Inferior in it's Measurement of Central Corneal Thickness Compared to the Ultrasound Pachymeter, Lenstar and Pentacam.
Brief Title: Assessment of the Occuity PM1 Pachymeter
Status: Completed | Type: Observational
Sponsor: Occuity Limited (Industry)
Collaborators: City, University of London (Other); Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ETH2021-1765
Record Dates: First submitted 2023-05-12; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Glaucoma Eye
Keywords: Cornea; Ocular; Glaucoma
MeSH Terms: conditions — Corneal Diseases; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Research Study: Is the Occuity pachymeter non inferior in it's measurement of central corneal thickness compared to the ultrasound pachymeter, Lenstar and Pentacam.

SUMMARY:
To determine whether the Occuity PM1 device is non-inferior in measuring central corneal thickness when compared to ultrasound pachymetry, the Lenstar and the Pentacam.

The Investigation aims to assess long-term safety of the Occuity PM1 device when used under the conditions and for the purposes intended, to ensure it will not compromise the clinical condition or the safety of patients, or the safety and health of users or, where applicable, other persons.

The central corneal thickness measurements taken by the three devices: Occuity PM1, the ultrasound pachymeter and Lenstar. Demonstrating that the Occuity PM1 Pachymeter is not inferior to the LenStar in terms of equivalency to a 95% confidence level using the Bland Altmen equation/approach based on +/-20micron equivalency.

The investigators would like to measure the thickness of the cornea, which is the clear window at the front of the eye. A corneal thickness measurement is important for several reasons. The measurement can tell an eye care professional if the cornea is swollen, which may mean the particiapnt have an increase in fluid within the cornea. Also, assessing corneal thickness can help in the diagnosis of glaucoma and the measurement is important if the participant is going to have eye surgery.

The instruments that are currently in use are usually very large and quite expensive and therefore not ideal for use as part of routine eye care. Some instruments require contact with the surface of the eye, which may be uncomfortable.

Occuity Ltd. is a medical device company based in Reading, which has been investigating this. They have developed a new instrument (called the 'PM1 Pachymeter') for measuring the thickness of the cornea. The instrument shines a harmless low power beam into the eye and then measures the light reflected back from the eye in order to check the thickness of the cornea. The low power beam is not a visible light and so the participant will not be able to see it. s study will assess how closely the eye measurements taken from the new PM1 Pachymeter matches eye measurements taken from two other devices that are currently on the market. The goal is to provide a non-contact, hand-held meter that is fast and easy to use without the need to contact the eye.

DETAILED DESCRIPTION:
The cornea is a thin, transparent structure at the front of the eye; its surface, as well as the overlying tear film, is responsible for the majority of the eye's refractive power.

Accurate and precise measurement of corneal thickness is important in the diagnosis and management of many ocular diseases. In particular, the central corneal thickness (CCT) measurement is a key parameter to consider when planning for procedures such as refractive surgery, and in the diagnosis of glaucoma.

Refractive error is the leading cause of reversible visual impairment worldwide; it is therefore unsurprising corrective refractive surgery is one of the most widely performed procedures globally. In the United Kingdom, the most frequently performed refractive surgery are laser assisted surgical procedures, such as laser assisted in situ keratomileusis (LASIK), Laser epithelial keratomileusis (LASEK), and Photorefractive Keratectomy (PRK). All of these techniques involve ablating the cornea with a laser to achieve a specific shape. Having an accurate measurement of corneal thickness is therefore of utmost importance in the planning stages, as excessive ablation of the cornea can lead to corneal ectasia, a significant complication of refractive surgery .

Glaucoma is a progressive disease which causes irreversible vision loss, and with ever aging populations, it is now one of the leading causes of irreversible blindness worldwide. Although it is considered to be multifactorial in aetiology, with both genetic and acquired factors contributing to its development and progressions, it is still widely accepted that the intraocular pressure (IOP) is the only modifiable factor in its management to prevent or slow further visual loss. (5).

IOP measurement is typically done in hospital clinics using a Goldmann applanation tonometer. The pressure reading is affected by the corneal thickness - a thick cornea will give a falsely elevated IOP reading, which may result in a patient with healthy eyes being commenced on unnecessary treatment, while conversely a thin cornea may give a falsely low pressure reading, which can result in patients with glaucoma not being started on sight-saving treatment. It has been estimated that a 10% increase in CCT can result in an apparent IOP increase of 3.4mmHg (2).

Ultrasound Pachymeter The ultrasound pachymeter (UP) is currently the gold standard method , as well as the most widely used to measure CCT. In comparative device studies, the ultrasound pachymeter has been shown to provide the most repeatable measurements . In addition, it is a small and portable handheld device, which makes it very convenient and timesaving to use during clinic appointments.

However, there are several negative aspects to the UP. First, it is necessary for the device to make direct contact with the cornea, which introduces the risk of corneal abrasions and subsequent infection. Second, anaesthetic eye drops need to be used for the patients to tolerate the corneal touch, and studies have shown that after instillation of anaesthetic eye drops, the CCT measurement is increased compared to before the use of anaesthetic, which can lead to a systematic over-reading of IOP. Third, the UP can be difficult to use, as it is necessary for the probe to contact the cornea perpendicularly, and exactly at the centre of the cornea to achieve the most accurate reading, which is difficult to achieve even with good staff training and experience. Lastly, despite the use of anaesthetic, measurement using this device is uncomfortable, and sometimes poorly tolerated due to the corneal touch, especially by the paediatric population.

While there are optical devices available on the market which can measure CCT without the instillation of anaesthetic or corneal touch, they tend to be bulky machines which are not portable and require specialist training to use. This makes their use in busy hospital clinics and community optometry practices less feasible.

There is a clear need to develop a device which can measure CCT accurately without necessitating corneal touch and use of topical anaesthetic, as well as being easily portable. There is no such device available on the market currently, and in our search in the clinical trial databases and Occuity did not identify any active trials investigating similar devices.

Occuity PM1 Pachymeter The Occuity device is a new handheld, non-contact, optical pachymeter, which utilise a low power, eye safe near infrared (1310nm) beam to measure the corneal thickness.

The device has an intuitive touchscreen display interface, and a series of 9 LEDs which provides the illumination needed to align the device in front of the eye. Once alignment is achieved, the measurement can take place by pressing the start button on the touchscreen display. During preliminary testing at the parent company, it has been shown the alignment and measurement process takes less than 10 seconds in total, after which a reading will be shown on the digital display of the device. The device is reported to have high reliability (variation of approximately 10um with repeat readings of the same eye), and comparable results to the Lenstar LS900 Biometer during initial testing.

The LED light system consist of a partial ring of 9 white LEDs at a radius of 8.75mm and spaced at 30° intervals. The total power is 2.4 mWm-2 which is will within the 10 mWm-2 blue light hazard eye safety limit. The maximum power of the infrared beam is 50µW, which given the expected exposure time of less than 10 seconds, is considered Class 1 eye safe according to BS EN 60825.

Lenstar LS 900 (Haag-Streit AG, Koeniz, Switzerland) The Lenstar is an optical device which utilises an 820mm super-luminescent diode and allows for high resolution measurements of the structures in the eye, including CCT. Its use is well established in the hospital clinic setting, and measurements do not require the use of anaesthetic drops or corneal touch. A drawback of this device is that it is large and heavy, and therefore not portable or as fast to use, unlike the ultrasound pachymeter or the Occuity PM1 device.

Pentacam (Oculus Optikgerate GmbH (Germany) Very similar to the Lenstar, the Pentacam is an optical device which also utilises an 820mm super-luminescent diode and allows for high resolution measurements of the structures in the eye, including CCT. Its use is well established in the hospital clinic setting, and measurements do not require the use of anaesthetic drops or corneal touch. A drawback of this device is that it is large and heavy, and therefore not portable or as fast to use, unlike the ultrasound pachymeter or the Occuity PM1 device.

ELIGIBILITY:
Inclusion Criteria:

The participant must meet ALL the following criteria to be considered eligible for the study:

* Male or Female, aged 18 years or above.
* Participant is willing and able to give informed consent for participation in the study.
* Able and willing to comply with all study requirements.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Any ocular surgery within 6 months
* Known active corneal abnormalities (e.g. Keratoconus, epithelial defects)
* Previous corrective refractive surgery (e.g. LASIK, PRK)
* Current ocular inflammatory or infectious disease (e.g. Uveitis, keratitis, corneal ulcers)
* Contact lens use within the last week
* Any contraindications to use of topical anaesthetic eye drops
* Any other pathology which the clinician or investigator believe may affect the accuracy of the CCT measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: United Kingdom
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
To determine whether the Occuity PM1 device is non-inferior in measuring central corneal thickness when compared to ultrasound pachymetry, the Lenstar and the Pentacam. | upto 3 months
  The central corneal thickness measurements taken by the three devices: Occuity PM1, the ultrasound pachymeter and Lenstar. Demonstrating that the Occuity PM1 Pachymeter is not inferior to the LenStar in terms of equivalency to a 95% confidence level using the Bland Altmen equation/approach.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrenson, Professor, Principal Investigator — City, University of London
Locations (1):
- Occuity Limited, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
A published paper will be submitted
Supporting Information: CSR
Time Frame: Draft copy is available now 19-APR-2023 and is under formal review

DOCUMENTS (1):
  • Study Protocol (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT05895617/Prot_000.pdf